CLINICAL TRIAL: NCT07215143
Title: Transcatheter Aortic Valve Implantation With Myval THV (OCTACOR/OCTAPRO) in Patients With a Failing Successfully Im-planted First Transcatheter Heart Valve
Brief Title: Observational Study to Collect Data of Patient Which Recieving a TAVI in TAVI Procedure
Acronym: REDO-TAVI
Status: Not yet recruiting | Type: Observational
Sponsor: IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Sponsor
Other Study IDs: BO-002
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with aortic valve stenosis often undergo transcatheter aortic valve implantation (TAVI) today. This biological valve can wear out or leak over time. In such cases, a second catheter-based procedure may be necessary, in which a new valve is inserted into the old one - a so-called TAVI-in-TAVI procedure. This method is considered a gentle alternative to repeat open heart surgery.

The trial will include around 300 patients from several European centres who are scheduled to undergo or have already undergone a TAVI-in-TAVI procedure with the Myval valve. Participation includes follow-up observation for a period of up to five years. Data collection will take place exclusively within the framework of regular medical care. This includes information on pre-existing conditions, the procedure, complications and subsequent hospital stays. Imaging examinations such as echocardiography or CT scans can also be centrally evaluated if they are performed routinely.

ELIGIBILITY:
Inclusion Criteria:

* A TAVI-in-TAVI procedure with implantation of the Myval THV (Oc-taCor/OctaPRO) into a previously implanted (≥3 months) failing transcatheter heart valve of any kind is either planned, has al-ready been performed, or was attempted, based on a clinical indi-cation established by the treating heart team.
* Age: 18 years or more
* Informed consent has been obtained.

Exclusion Criteria:

* Participation in an interventional clinical trial
* Limited life expectancy <12 months
* Foreseeable problems in performing follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffers from aortic valve stenosis due to an failure of a previous implanted aortic valve.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2033-01 (Estimated); Study Completion 2033-06 (Estimated)

PRIMARY OUTCOMES:
VARC-3 (Valve Academic Research Consortium Version 3)) | at 30 days

IPD SHARING:
Plan to Share IPD: No